CLINICAL TRIAL: NCT05142748
Title: Study of Pulmonary Infections (Pneumonia) in Kidney Transplant Recipients Admitted to Hospital
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2021Ao001
Record Dates: First submitted 2021-11-17; First posted 2021-12-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Kidney Transplant Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to identify prognosis factors associated with in-hospital complications and assess the epidemiology, management, and outcomes of community-acquired pneumonia in a kidney transplant recipients' cohort. The investigators intend to identify each stay by a national database. Then they will be consulted by 2 clinicians to assert CAP clinical definition. After that radiographic evidence will be reviewed to validate CAP diagnoses. Then clinical data are collected in each center.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients
* at least 18 years
* admitted to hospital for CAP. Non-inclusion criteria were:

Exclusion Criteria:

* incomplete CAP definition
* hospital-acquired pneumonia
* another diagnosis explaining the symptoms
* patients with non-functional kidney graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
In-hospital complications | inhospital stay, an average of 30 days
  In-hospital death, transfer to intensive care units (ICU) and prolonged stays

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided